CLINICAL TRIAL: NCT05014659
Title: The Impact of Creatine Supplementation on Vascular Endothelial Function, Blood Flow and Functional Exercise Capacity
Brief Title: Creatine Monohydrate Supplementation and Vascular Endothelial Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida State University (Other)
Responsible Party: Principal Investigator, Holly Clarke, Principle Investigator, Florida State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00000764
Record Dates: First submitted 2021-08-19; First posted 2021-08-20 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Endothelial Dysfunction; Oxidative Stress
Keywords: Older adults; Flow mediated dilation
MeSH Terms: interventions — Creatine; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Creatine monohydrate (Experimental): Participants received 4 x 5g doses of creatine monohydrate (powdered form) for 5 days, followed by 1 x 5g doses of creatine monohydrate (powdered form) for 23 days.
  Interventions: Dietary Supplement: Creatine monohydrate
- Placebo (Placebo Comparator): Participants received 4 x 5g doses of placebo (powdered Maltodextrin) for 5 days, followed by 1 x 5g doses of placebo (powdered Maltodextrin) for 23 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Creatine monohydrate — 4 x 5g doses daily for 5 days, followed by 1 x 5g dose daily for 23 days.
  Arms: Creatine monohydrate
Dietary Supplement: Placebo — 4 x 5g doses daily for 5 days, followed by 1 x 5g dose daily for 23 days.
  Other Names: Maltodextrin
  Arms: Placebo

SUMMARY:
To determine the effects of 4 weeks of creatine monohydrate supplementation on markers of macrovascular and microvascular function, cognitive performance, and physical performance.

DETAILED DESCRIPTION:
This is a randomized, double-blind (participant and principle investigator), placebo-controlled, crossover study.

After a pre-screen telephone interview, potential participants will be invited to Florida State University for a "Screening visit". During this visit, individuals will be provided with a verbal and written explanation of the study. Individuals will complete an informed consent, a health history questionnaire and physical activity readiness questionnaire. If they meet study inclusion criteria, they will undergo anthropometric measurements and a venous blood draw to determine cardiovascular and kidney disease risk profile. If cleared for participation, participants will be asked to complete a "3-Day Food Log" prior to their next visit.

Once qualified, participants will return to the laboratory to undergo their "Baseline Testing Visit". Following the completion of the first "Baseline Testing Visit", participants will be randomly assigned to one of two interventions: 1) creatine monohydrate; or, 2) maltodextrin "placebo". Participants will be given their supplement and asked to complete the supplementation protocol, complying with instructions given. Following the 4-week supplementation period, participants will return to the laboratory for their "Post-Supplement #1 Testing". During this visit, all procedures from the "Baseline Testing Visit" will be repeated.

Once these measurements are completed, participants will be asked to return to their normal daily lifestyles for a 4-week "wash-out" period. During these 4-weeks, participants will be contacted weekly to ensure retention and to schedule the next visit. Following the washout, participants will return to the laboratory to undergo another "Baseline Testing Visit", completing the exact procedures as outlined previously. Following this, participants will be given their remaining supplement intervention. Following the intervention, participants will return to the lab for their final "Post-Supplement #2 Testing" to conclude the study.

ELIGIBILITY:
Inclusion Criteria:

* both male and female
* 50-64 years old
* no restrictions based on race, ethnicity, or socioeconomic status
* sedentary individuals (<20 minutes; <3 days/wk. physical activity)
* post-menopausal women (has experienced 12 consecutive months without menstruation for >5 years).

Exclusion Criteria:

* <50 or ≥65 years of age
* Subjects participating in regular exercise (>20 min/day, >3 days/week)
* female subjects who are pregnant, lactating or 1 month post-partum
* currently consuming or had consumed creatine supplementation <1 month prior to screening
* currently consuming or consumed nitric oxide supplementation <1 month prior to screening
* currently consuming or had consumed Vitamin C supplementation <2 weeks prior to screening
* individuals who report chronic infections
* individuals reporting paralysis due to stroke
* individuals reporting advanced Parkinson's disease
* individuals reporting severe rheumatoid arthritis or other serious orthopedic problems that would prevent performance of the exercise tasks
* individuals currently taking medications that may affect central or peripheral circulation
* individuals with known cardiovascular and/or metabolic disease
* current smokers or those who quit <6 months prior to screening
* individuals with hypercholesterolemia (total cholesterol > 200mg/dL, high density lipoprotein <40 mg/dL, low density lipoprotein >130mg/dL)
* individuals with hypertension (systolic blood pressure > 150 mmHg and/or diastolic blood pressure >95mmHg).
* individuals with known kidney disease
* individuals with known liver disease

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-10-17 (Actual); Primary Completion 2022-12-12 (Actual); Study Completion 2022-12-12 (Actual)

PRIMARY OUTCOMES:
Change from baseline in brachial artery flow mediated dilation (FMD%) at week 4 | Baseline and Week 4
  FMD% is a validated, non-invasive, standardized method of measuring the ability of an artery to respond to a stimulated increase in blood flow via vasodilation. Increase in blood flow will be stimulated by inflating a forearm cuff for 5 minutes, then rapidly releasing this cuff. Brachial artery in the participants right arm will be identified/imaged using a Philips Doppler Ultrasound. Resting diameter will be measured in millimeters, and max dilation will be the maximum diameter in millimeters following increased blood flow (cuff release). FMD% will be calculated by [(max diameter - resting diameter) / resting diameter] x 100.
  Change = Week 4 Score - Baseline Score
Change from baseline in forearm microvascular reperfusion rate (%/sec) at week 4 | Baseline and Week 4
  Microvascular reperfusion rate will be assessed using a near-infrared spectroscopy (NIRS) unit placed on the forearm during the FMD assessment. This small, non-invasive NIRS unit will allow for the determination of forearm muscle tissue oxygen saturation during FMD. The microvascular reperfusion rate (%/sec) will be determined by analyzing the upward slope of tissue saturation following FMD cuff release.
  Change = Week 4 Score - Baseline Score
Change from baseline in brachial-ankle pulse wave velocity (baPWV) at week 4 | Baseline and Week 4
  PWV is a validated, non-invasive, clinical technique used to measure arterial stiffness. Participants will lay supine, and 4 blood pressure cuffs will be wrapped around the limbs. One cuff on each arm (brachial artery) and one cuff on each ankle (posterior tibial artery). The distance between the two sampling points (arms and ankles) will be calculated according to the height of the subject. PWV is measured as the distance between two recording sites divided by the transit time of the pulse wave detected. PWV will be given as meters/second.
  Change = Week 4 Score - Baseline Score
Change from baseline in augmentation (AUG) and augmentation index (AIx) using pulse wave analysis (PWA) at week 4 | Baseline and Week 4
  Both AUG and AIx are determined based on waveforms captured using a pulse wave analysis device (PWA). PWA is a validated, non-invasive technique used to determine central arterial stiffness via the assessment of the radial pulse (wrist). PWA will be measured using a tonometer which is gently pressed against the radial pulse point. Ten seconds of high-quality waveforms will be captured and analyzed to determine AUG (the pressure added to the forward wave by the reflected wave; measured in mmHg) and AIx (a measure of the effect of the wave reflection on the second systolic peak; expressed as a %).
  Change = Week 4 Score - Baseline Score
Change from baseline in oxidized low density lipoprotein (oxLDL) at week 4 | Baseline and Week 4
  OxLDL is a commonly used, validated, blood biomarker of lipid oxidation. OxLDL is thereby indicative of oxidative stress. A small amount of venous blood will be drawn (~5ml) at the beginning of every visit, centrifuged, and then stored in a -80 freezer. Plasma will later be used to analyze levels of OxLDL using a commercially available enzyme-linked immunoassay.
  Change = Week 4 Score - Baseline Score
Change from baseline in tetrahydrobiopterin (BH4) at week 4 | Baseline and Week 4
  BH4 is a very important cofactor necessary for the natural production of nitric oxide - a substance produced by the body and majorly responsible for the vasodilation (increase in diameter) of major arteries, such as the brachial artery. BH4 has been shown to decrease with age and with higher levels of systemic oxidative stress. A small amount of venous blood will be drawn (~5ml) at the beginning of every visit, centrifuged, and then stored in a -80 freezer. Plasma will then later be used to analyze levels of BH4 using a commercially available enzyme-linked immunoassay.
  Change = Week 4 Score - Baseline Score
Change from baseline in malondialdehyde (MDA) at week 4 | Baseline and Week 4
  MDA is a commonly used, validated, blood biomarker of oxidative stress. A small amount of venous blood will be drawn (~5ml) at the beginning of every visit, centrifuged, and then stored in a -80 freezer. Plasma will then later be used to analyze levels of MDA using a commercially available enzyme-linked immunoassay.
  Change = Week 4 Score - Baseline Score
Change from baseline in total 6-minute walking distance (6MWT) at week 4 | Baseline and Week 4
  The 6 minute walk test (6MWT) assesses distance walked over 6 minutes as a sub-maximal test of aerobic capacity/endurance. The participant will be asked to walk on a pre-measured track for a total of 6 minutes, and total distance covered will be measured in meters following completion.
  Change = Week 4 Score - Baseline Score
Change from baseline in total torque produced (total Nm) per set at week 4 | Baseline and Week 4
  In order to assess physical performance, participants will perform right knee extension and flexion for a total of 3 sets, each consisting of 30 repetitions, with 1 minute recovery between each set. This assessment will be carried out on a Biodex Isokinetic Dynamometer, which will track force produced in Newton meters (Nm) for each repetition. For each individual set, the peak torque of each repetition will be summed, and this value will be used to represent isokinetic performance. This data will be presented as total newton-meters (Nm) produced per set.
  Change = Week 4 Set 1 Score - Baseline Set 1 Score Week 4 Set 2 Score - Baseline Set 2 Score Week 4 Set 3 Score - Baseline Set 3 Score
Change from baseline in time taken to complete (seconds) the Trail Making Test (TMT) at Week 4 | Baseline and Week 4
  The TMT is a measurement of visual attention and task switching and has been validated for its use in neuropsychological assessment. Both parts of the TMT (Part A + Part B) consist of 25 circles distributed over a sheet of white paper. In Part A of the TMT, circles are numbered 1 - 25, and the participant will be instructed to connect numbers consecutively in ascending order (ex. 1,2,3,4…). In Part B of the TMT, circles include both numbers (1 - 13) and letters (A - L). Participants will also be asked to draw lines to connect these circles in an ascending manner, but with the added task of alternating between numbers and letters (ex. 1-A-2-B-3-C…). During both trials the participant will be asked to connect the circles as quickly as possible. Time taken to complete each trial (Part A + Part B) will be recorded (seconds).
  Change = Week 4 Score - Baseline Score
Change from baseline in maximum number recall (#) achieved in the Digit Span memory recall test at Week 4 | Baseline and Week 4
  A digit span (DS) memory recall test will be used to assess short-term memory. Both forward and backward DS testing remains one of the most widely utilized neuropsychological tests used to assess short-term verbal memory. Participants will complete both a forward-DS (FDS) and a backward-DS (BDS) test. Participants will be read a sequence of numbers at a rate of 1 digit/second, in a monotonous and clear tone. Each sequence will vary in length, from 2 numbers to 9 numbers. Participants will have 2 attempts to successfully repeat the sequence of numbers. The test will be discontinued after the failure to repeat a sequence on both attempts. Following this, participants will complete a BDS. Numbers will now have to be repeated backwards by the participant. Both digit span tests will be scored and reported separately as "span scores" (the maximum number of digits correctly produced forward or backwards by the participant).
  Change = Week 4 Score - Baseline Score

SECONDARY OUTCOMES:
Change from baseline in body fat percent (BF%) at week 4 | Baseline and Week 4
  Body fat %, or the percent of an individuals body weight that is fat mass, will be determined using a dual-energy X-ray absorptiometry (DXA) scan. Participants will lay supine on the DXA table, and be scanned from head to toe. This procedure involves a minimal amount of radiation that is within an acceptable range. The amount of radiations per scan is less than one tenth of the amount used during a normal chest x-ray and equivalent to one day of exposure to natural background radiation. The amount of radiation used during a DXA scan is considered safe for adults. BF% will then be determined by the DXA computer software.
  Change = Week 4 Score - Baseline Score
Change from baseline in body lean mass (grams) at week 4 | Baseline and Week 4
  Lean mass, or the amount in grams of an individuals body weight that is composed of lean tissue such as muscle, will be determined using a dual-energy X-ray absorptiometry (DXA) scan. Participants will lay supine on the DXA table, and be scanned from head to toe. This procedure involves a minimal amount of radiation that is within an acceptable range. The amount of radiations per scan is less than one tenth of the amount used during a normal chest x-ray and equivalent to one day of exposure to natural background radiation. The amount of radiation used during a DXA scan is considered safe for adults. Lean mass (g) will then be determined by the DXA computer software.
  Change = Week 4 Score - Baseline Score
Change from baseline in body fat mass (grams) at week 4 | Baseline and Week 4
  Fat mass, or the amount in grams of an individuals body weight that is composed of fat tissue such as visceral fat, will be determined using a dual-energy X-ray absorptiometry (DXA) scan. Participants will lay supine on the DXA table, and be scanned from head to toe. This procedure involves a minimal amount of radiation that is within an acceptable range. The amount of radiations per scan is less than one tenth of the amount used during a normal chest x-ray and equivalent to one day of exposure to natural background radiation. The amount of radiation used during a DXA scan is considered safe for adults. Fat mass (g) will then be determined by the DXA computer software.
  Change = Week 4 Score - Baseline Score
Change from baseline in total body water (liters) at week 4 | Baseline and Week 4
  The total amount of body water will be determined by using a Bioelectrical Impedance Analysis device (BIS). BIS works by having subjects lay supine whilst electrodes are placed on both the right ankle and right wrist. A low level, imperceptible electrical current is then sent through the body, travelling from electrode A to electrode B. The flow of the current is affected by the amount of water in the body; therefore the BIS can estimate how much water is present in the body (liters). Furthermore, this total amount will then be categorized as either intracellular fluid (fluid found within cells) or extracellular fluid (fluid found outside cells). This BIS will be used to measure any possible fluids shifts.
  Change = Week 4 Score - Baseline Score
Change from baseline in resting systolic blood pressure (mmHg) at week 4 | Baseline and Week 4
  Resting systolic blood pressure will be measured following 10 minutes of laying supine in a temperature controlled, dimly lit room, using a commercially available automatic blood pressure device (Omron).
  Change = Week 4 Score - Baseline
Change from baseline in resting diastolic blood pressure (mmHg) at week 4 | Baseline and Week 4
  Resting diastolic blood pressure will be measured following 10 minutes of laying supine in a temperature controlled, dimly lit room, using a commercially available automatic blood pressure device (Omron).
  Change = Week 4 Score - Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Holly E Clarke, PhD, Principal Investigator — Florida State University
Locations (1):
- Sandels Building, Tallahassee, Florida, United States

IPD SHARING:
Plan to Share IPD: No
Participant data will not be shared with anyone who is not an approved research team member, as indicated in this study's Florida State University Institutional Review Board document.